CLINICAL TRIAL: NCT03166007
Title: Abdominal Massage for Neurogenic Bowel Dysfunction in People With Multiple Sclerosis (AMBER Abdominal Massage for Bowel Dysfunction Effectiveness Research).
Brief Title: Abdominal Massage for Bowel Dysfunction
Acronym: AMBER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/127
Record Dates: First submitted 2016-05-25; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Neurogenic Bowel Dysfunction; Abdominal massage
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimised bowel care + abdominal massage (Experimental): In addition to optimised bowel care as described below for the control group, the Intervention Nurse will teach the participant and/or their carer in the intervention arm how to deliver the abdominal massage. This will include viewing the massage DVD and the abdominal massage training booklet, as well as the demonstration of the technique on the participant by the Intervention Nurse.
  Interventions: Behavioral: Abdominal massage; Behavioral: Optimised bowel care
- Optimised bowel care (Active Comparator): During a 1 hour outpatient appointment, the participants' existing bowel care routine will be reviewed and optimised. For example, explaining the necessity of adequate fluid intake. No change in medication will be advocated.
  Interventions: Behavioral: Optimised bowel care

INTERVENTIONS:
Behavioral: Abdominal massage — The participant should be supine and in a relaxed atmosphere, though this may depend on level of disability. The massage comprises 4 basic strokes (10minutes); Stroking from the small of the back over the iliac crest and down both sides of the pelvis towards the groin; Effleurage follows the direction of the ascending colon across the transverse colon and down the descending colon. This is repeated several times with increasing pressure; Palmar kneading tracks down the descending colon up the ascending colon and down the descending colon once again. Effleurage is repeated and continued with a relaxing transverse stroke over the abdomen; Vibration over the abdominal wall to relieve flatus concludes the massage session. The participants in this group will receive one telephone call per week for 6 weeks and again at 24 weeks to further discuss their bowel management.
  Arms: Optimised bowel care + abdominal massage
Behavioral: Optimised bowel care — During a 1 hour outpatient appointment, the participants' existing bowel care routine will be reviewed and optimised. For example, explaining the necessity of adequate fluid intake. No change in medication will be advocated. The participants in this group will also receive one telephone call per week during the following 6 week period to further discuss their bowel management and again at 24 week time point.

SUMMARY:
The aim of the AMBER trial is to determine the effectiveness and cost effectiveness of abdominal massage as part of the adjunct to bowel care in people with Multiple Sclerosis who have problems with their bowel i.e. faecal incontinence and/or constipation.

DETAILED DESCRIPTION:
Neurogenic bowel dysfunction (NBD: constipation and/or faecal incontinence) is common in people with multiple sclerosis (MS) and is rated as the most severe impact of their disease/injury, above wheelchair dependence. Despite this, current treatment options are limited, poorly evaluated and complex.

This research aims to find out whether abdominal massage can help improve the symptoms of NBD in these patients. A small study has already shown that it is possible for patients or carers to perform abdominal massage and in some cases this helped the patient with their symptoms. A larger study is now required to confirm the results one way or another.

Patients with Multiple Sclerosis who attend one of the participating study centres who are bothered by constipation and or faecal incontinence will be asked to take part if they fit the other requirements for the trial. Those who agree to take part will be allocated at random to one of two groups, one will receive advice on the management of bowel dysfunction (called optimised bowel care), and the other will receive the same advice and will be taught how to do the abdominal massage (called abdominal massage and optimised bowel care). Both groups will visit a specialist nurse for 1 additional hour after their normal clinical appointment, or at an agreed time, to receive optimised bowel care advice. The patients in the intervention group +/or their carers will receive training on abdominal massage and a DVD/copy of demonstration of the massage for home use. All patients will also be called weekly for 6 weeks to discuss their bowel care.

The investigators will measure the results of treatment after 6 and 24 weeks. The investigators are primarily interested in whether patients in the intervention group (receiving optimized bowel care & abdominal massage) have had more of an improvement in their NBD score at 24 weeks after they start the study that the control group (receiving optimized bowel care only). The investigators also want to find out how bad the constipation and bowel symptoms are, how much this affects their life and if they have any problems with their bladder. The investigators will also measure the costs of the treatments and any costs to the patient and their family, and balance these against any benefits of the intervention treatment.

During the trial the investigators will assess how well the optimized bowel care and abdominal massage training was delivered by speaking with nurses and listening to recordings of some of the telephone calls. The investigators will talk to the patients to find how they perceive the treatment they received and how they got on during the treatment period and once the treatment finished. The investigators will explore how the treatment delivery and patient's perceptions impact on the patients NBD symptoms.

The investigators have worked out from previous research that if 200 patients take part and most complete the trial, there will be enough data to successfully compare the treatments to find out if one is better than the other. Individual participation will be entirely voluntary and the investigators do not believe there are any risks associated with taking part.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 18 years;
* Diagnosis of MS (in a stable phase i.e. no MS relapse for 3 months);
* No major change of medication for 1 month e.g. introduction of disease modifying medications;
* Individual is bothered by their bowel dysfunction, and;
* Must not have used abdominal massage for at least 2 months.

Exclusion Criteria:

* Individuals who are unable to undertake the massage themselves or do not have a carer willing to do it;
* Individuals who are unable to understand the study processes;
* Individuals who have contraindications to abdominal massage e.g. history of abdominal/pelvic cancer, hiatus, inguinal or umbilical hernia, rectal prolapse, Inflammatory Bowel Disease, pregnancy and past history of volvulus.
* Recent abdominal scars, abdominal wounds or skin disorders that may make abdominal massage uncomfortable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2014-06; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 24 weeks Neurogenic Bowel Dysfunction Score (NBDs) | Baseline - 24 weeks
  NBDs is a 10 item questionnaire covering frequency of bowel movements, headache, perspiration or discomfort during defecation; medication for constipation or faecal incontinence; time spent on defecation; frequency of digital stimulation or evacuation; frequency of faecal incontinence; flatus incontinence; and perianal skin problems. Maximum score is 47 with over 14 considered severe.

SECONDARY OUTCOMES:
Neurogenic Bowel Dysfunction Questionnaire (NBD PROM) - change in Score from Baseline to 24 weeks | Baseline - 24 weeks
Constipation Symptoms (Constipation Scoring System (CSS)) - change in Score from Baseline to 24 weeks | Baseline - 24 weeks
Bowel Symptoms (7 day diary) - change in Score from Baseline to 24 weeks | Baseline - 24 weeks
Radio Opaque Marker transit tests - change in Score from Baseline to 24 weeks | Baseline - 24 weeks
  One Site only
Adherence to massage schedule (7 day diary) - change in Score from Baseline to 24 weeks | Baseline - 24 weeks
  Intervention arm only
Bladder Function (Qualiveen Questionnaire Short Form) - change in Score from Baseline to 24 weeks | Baseline - 24 weeks
Health Status (EQ-5D-5L Health Questionnaire) - change in Score from Baseline to 24 weeks | Baseline - 24 weeks
Change of medication (Concomitant Medication Form) | Over the study duration (24 weeks)
Patient Resource Questionnaire - cost and use of NHS services (£) | Baseline, 1-6weeks, 12 weeks, 18 weeks and 24 weeks
Patient Resource Questionnaire - cost to the patients and their families/carers (£) | Baseline, 1-6weeks, 12 weeks, 18 weeks and 24 weeks
Patient Resource Questionnaire - incremental costs, QALYs and incremental cost per QALY derived by the economic model (£) | Baseline, 1-6weeks, 12 weeks, 18 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Doreen McClurg, Principal Investigator — Glasgow Caledonian University
Locations (1):
- Glasgow Caledonian University - NMAHP RU, Glasgow, Glasgow City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Results will be published, lay summaries produced and massage training guidelines (+DVD) will be made available.

REFERENCES:
- [Derived] Todd CL, Johnson EE, Stewart F, Wallace SA, Bryant A, Woodward S, Norton C. Conservative, physical and surgical interventions for managing faecal incontinence and constipation in adults with central neurological diseases. Cochrane Database Syst Rev. 2024 Oct 29;10(10):CD002115. doi: 10.1002/14651858.CD002115.pub6. PMID 39470206
- [Derived] McClurg D, Harris F, Goodman K, Doran S, Hagen S, Treweek S, Norton C, Coggrave M, Norrie J, Rauchhaus P, Donnan P, Emmanuel A, Manoukian S, Mason H. Abdominal massage plus advice, compared with advice only, for neurogenic bowel dysfunction in MS: a RCT. Health Technol Assess. 2018 Oct;22(58):1-134. doi: 10.3310/hta22580. PMID 30375324